CLINICAL TRIAL: NCT04652687
Title: VIA Disc NP Registry
Status: Terminated | Type: Observational
Why Stopped: Sponsor decision.
Sponsor: VIVEX Biologics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: VIV-001-020
Record Dates: First submitted 2020-11-03; First posted 2020-12-03 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Discogenic Pain; Back Pain; Back Pain, Low
Keywords: back pain
MeSH Terms: conditions — Back Pain; Low Back Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- VIA Disc NP: Patients meeting study criteria receiving Vivex VIA Disc NP injection as treatment
  Interventions: Other: VIA Disc NP (HCT/P)

INTERVENTIONS:
Other: VIA Disc NP (HCT/P) — VIA Disc NP - Allograft tissue injection

SUMMARY:
Registry is to observe and trend patterns of care and outcomes for patients treated with VIA Disc NP.

DETAILED DESCRIPTION:
The Registry is intended to collect data for patients having received treatment with VIA Disc NP.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Understand and sign the informed consent form (as applicable)
* VIA Disc NP injection is scheduled for 1 or more levels

Exclusion Criteria:

* VIA Disc NP injection is not performed

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Registry will include at least 10,000 patients diagnosed with and treated for back pain across approximately 200 selected sites.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2020-05-03 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
Patient self-reporting of daily function | 1, 3, 6, 12, 24, & 36 months
  Change in scores from Oswestry Disability Index (ODI). An index comprising of ten categories of function to quantify disability due to back pain.
Patient self-reported back pain | 1, 3, 6, 12, 24, & 36 months
  Change in Numeric Rating Scale (NRS) scores. Eleven point pain scale used for patient self-reporting of back pain, which ranges from 0 (no pain) to 10 (the worst pain imaginable).

SECONDARY OUTCOMES:
Patient self-reported mental health | 1, 3, 6, 12, 24, & 36 months
  Change in patient reported anxiety and depression scores. Four question scale used for patient self-reporting of anxiety and depression which ranges from 0-2 (normal), mild (3-5), moderate (6-8), and severe (9-12).
Resource Utilization | 1, 3, 6, 12, 24, & 36 months
  Patient reported assessment of healthcare and resources utilized questions to treat ongoing back pain post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Finstein, MHA, Study Director — Vivex Biologics
Locations (32):
- United States (32):
  - Gateway Pain Solutions, Mesa, Arizona
  - Source Healthcare, Santa Monica, California
  - Interventional Pain Management, Walnut Creek, California
  - MD Pain, Englewood, Colorado
  - Western Rockies Interventional Pain Specialists, Grand Junction, Colorado
  - The Denver Spine & Pain Institute, Greenwood Village, Colorado
  - International Spine, Pain & Performance Center, Washington D.C., District of Columbia
  - The Orthopedic Institute, Gainesville, Florida
  - Southwest Florida Pain Center, Port Charlotte, Florida
  - FAST MD, Tampa, Florida
  - Florida Spine & Pain Specialists, Tampa, Florida
  - Florida Pain Medicine, Wesley Chapel, Florida
  - Orthopaedic Research Foundation, Indianapolis, Indiana
  - Anesthesiology & Pain Consultants, Lafayette, Louisiana
  - Interventional Pain Specialists, Opelousas, Louisiana
  - Michigan Interventional Pain Center, Brownstown, Michigan
  - Forest Health, Ypsilanti, Michigan
  - Nevada Advanced Pain Specialists, Reno, Nevada
  - Ainsworth Institute of Pain Management, New York, New York
  - Premier Pain Solutions, Asheville, North Carolina
  - Crystal Coast Pain Management, New Bern, North Carolina
  - Premier Pain, Loveland, Ohio
  - Invictus Healthcare System, Tulsa, Oklahoma
  - Center for Interventional Pain Spine, Chadds Ford, Pennsylvania
  - Atlantic Coast Pain Management, Conway, South Carolina
  - Southeastern Spine Institute, Mt. Pleasant, South Carolina
  - Specialist in Pain Management, Chattanooga, Tennessee
  - Vertex Spine, Franklin, Tennessee
  - Ortho Spine Surgery Institute, North Richland Hills, Texas
  - MD SpineCare and DC Medical Solutions, San Antonio, Texas
  - Advanced Spine and Pain Center, San Antonio, Texas
  - The Sprintz Center for Pain, Shenandoah, Texas

IPD SHARING:
Plan to Share IPD: No